CLINICAL TRIAL: NCT01438385
Title: Endoscopic Retrograde Cholangiopancreatography, Endoscopic Ultrasound and Interventional Endoscopy in Pancreatico-biliary, Gastrointestinal and Esophageal Disorders
Brief Title: Interventional Endoscopy Database for Pancreatico-biliary, Gastrointestinal and Esophageal Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief, Advanced Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1104011642
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Ampullary Cancer; Duodenal Cancer; Bile Duct Cancer; Bile Duct Disorders; Gallstones; Obstructive Jaundice; Pancreatic Disorders (Noncancerous); Colorectal Cancer; Esophageal Cancer; Barrett's Esophagus; Gastric Malignancies; Pancreatic Cancer; Pediatric Gastroenterology; Cholangiocarcinoma; Pancreatic Pseudocysts; Acute and Chronic Pancreatitis; Recurrent Pancreatitis; Cholangitis; Bile Leak; Biliary Strictures; Pancreatic Divisum; Biliary and Pancreatic Stones; Choledocholithiasis
Keywords: Pancreatico-biliary; Biliary; Bile Duct; Gastrointestinal disorder; Esophageal disorder
MeSH Terms: conditions — Duodenal Neoplasms; Bile Duct Neoplasms; Bile Duct Diseases; Gallstones; Jaundice, Obstructive; Pancreatic Diseases; Colorectal Neoplasms; Esophageal Neoplasms; Barrett Esophagus; Pancreatic Neoplasms; Cholangiocarcinoma; Pancreatic Pseudocyst; Pancreatitis, Chronic; Cholangitis; Pancreas Divisum; Choledocholithiasis; Gastrointestinal Diseases; Esophageal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interventional Endoscopy: Any group that went Interventional Endoscopy procedures.
  Interventions: Procedure: Interventional Endoscopy

INTERVENTIONS:
Procedure: Interventional Endoscopy — Advanced imaging endoscopic or therapeutic endoscopy
  Other Names: Advanced Endoscopy

SUMMARY:
Our institution performs therapeutic ERCP (Endoscopic retrograde cholangiopancreatography ), Endoscopic Ultrasound (EUS) and Interventional Endoscopy in around 1000 patients a year. Procedures such as biliary and/or pancreatic sphincterotomy, stents placement (metallic or plastic) and removal for revision, cysts and pseudocysts drainage are conducted in patients suffering from pancreatico-biliary disorders, gastrointestinal disorders and esophageal disorders. The investigators would like to assess prospectively the efficacy and safety of these routine procedures to permit identification of technical details about the procedures or other factors which might be associated with outcome or results. Assessment of these details would help us with problem identification and recommendations to improve health outcomes and quality of life in these patients.

DETAILED DESCRIPTION:
Our institution performs therapeutic ERCP (Endoscopic retrograde cholangiopancreatography ), Endoscopic Ultrasound (EUS) and Interventional Endoscopy in around 1000 patients a year. Procedures such as biliary and/or pancreatic sphincterotomy, stents placement (metallic or plastic) and removal for revision, cysts and pseudocysts drainage are conducted in patients suffering from pancreatico-biliary disorders, gastrointestinal disorders and esophageal disorders. The investigators would like to assess prospectively the efficacy and safety of these routine procedures to permit identification of technical details about the procedures or other factors which might be associated with outcome or results. Assessment of these details would help us with problem identification and recommendations to improve health outcomes and quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Any subject that underwent Interventional Endoscopy for Pancreatico-biliary, Gastrointestinal or Esophageal disorders.
* Above the age of 18 years

Exclusion Criteria:

* Any group that did not undergo Interventional Endoscopy for Pancreatico-biliary, Gastrointestinal or Esophageal disorders.
* Below the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any subject that underwent Interventional Endoscopy for Pancreatico-biliary, Gastrointestinal or Esophageal disorders.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2011-07; Primary Completion 2017-12-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Establishing a database that contains all Interventional Endoscopies | 5 years
  Collection of procedure specific details of all Interventional Endoscopies

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD Sharing

REFERENCES:
- [Derived] Tyberg A, Desai AP, Kumta NA, Brown E, Gaidhane M, Sharaiha RZ, Kahaleh M. EUS-guided biliary drainage after failed ERCP: a novel algorithm individualized based on patient anatomy. Gastrointest Endosc. 2016 Dec;84(6):941-946. doi: 10.1016/j.gie.2016.05.035. Epub 2016 May 26. PMID 27237786
- [Derived] Desai AP, Tyberg A, Kedia P, Smith MS, Martinez G, Zamarripa F, Schneider Y, Bertani H, Frazzoni M, Casas F, Khanna LG, Lambroza A, Kumta NA, Khan A, Sharaiha RZ, Salgado S, Gaidhane M, Sethi A, Kahaleh M. Optical coherence tomography (OCT) prior to peroral endoscopic myotomy (POEM) reduces procedural time and bleeding: a multicenter international collaborative study. Surg Endosc. 2016 Nov;30(11):5126-5133. doi: 10.1007/s00464-016-4859-0. Epub 2016 Apr 8. PMID 27059973